CLINICAL TRIAL: NCT00523185
Title: A Comparison of Lorazepam and Diazepam in the Treatment of Alcohol Withdrawal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 77757
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Last update posted 2007-08-31 (Estimated); Status verified 2007-08

CONDITIONS: Alcohol Withdrawal
Keywords: alcohol withdrawal; lorazepam; diazepam
MeSH Terms: interventions — Lorazepam; Diazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator)
  Interventions: Drug: Diazepam
- 1 (Active Comparator)
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Lorazepam — Lorazepam 1 to 2 mg by mouth or intravenously every two hours as needed for alcohol withdrawal symptoms.
  Other Names: Ativan
  Arms: 1
Drug: Diazepam — Diazepam 20 mg by mouth every two hours x 3 doses, or for parenteral treatment, diazepam 10 mg intravenously every one hour x 6 doses. Give additional diazepam 10 mg by mouth or intravenously every two hours as needed for alcohol withdrawal symptoms.
  Other Names: Valium
  Arms: 2

SUMMARY:
The purpose of this study is to compare the efficacy of two commonly used medications in the treatment of alcohol withdrawal, diazepam and lorazepam.

DETAILED DESCRIPTION:
Despite the frequent use of benzodiazepines for the treatment of alcohol withdrawal, studies comparing the efficacy of long and short half-life benzodiazepines in the treatment of alcohol withdrawal have shown mixed results. Due to the conflicting nature of published reports, clinicians have no clear indication as to which type of agent is preferable. The purpose of this study is to compare the efficacy of two commonly accepted medications in the treatment of alcohol withdrawal, diazepam and lorazepam, which are long and short half-life benzodiazepines, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of alcohol withdrawal
* History of alcohol use within 24 hours
* Ability to consent to participate in the study

Exclusion Criteria:

* Unwillingness to participate in the study
* Active abuse of other CNS depressants
* Acute intoxication with a CNS activating agent
* Severe hepatic dysfunction
* Pregnancy
* History of dementia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2003-05; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures include serial measures of vital signs and scores on the Clinical Institute Withdrawal Assessment for Alcohol-Revised scale (CIWA-Ar), a widely used scale that monitors alcohol withdrawal symptoms. | one to two weeks

SECONDARY OUTCOMES:
Secondary outcome measures include total benzodiazepine use. | one to two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Maldonado, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Palo Alto Veterans Affairs Hospital System, Palo Alto, California
  - Stanford Hospital and Clinics, Stanford, California

REFERENCES:
- [Derived] Maldonado JR, Nguyen LH, Schader EM, Brooks JO 3rd. Benzodiazepine loading versus symptom-triggered treatment of alcohol withdrawal: a prospective, randomized clinical trial. Gen Hosp Psychiatry. 2012 Nov-Dec;34(6):611-7. doi: 10.1016/j.genhosppsych.2012.06.016. Epub 2012 Aug 13. PMID 22898443